CLINICAL TRIAL: NCT03030651
Title: Effect of Breastfeeding Education and Support Intervention on Timely Initiation and Exclusive Breastfeeding in Southwest Ethiopia: a Cluster Randomized Controlled Trial.
Brief Title: Effect of Breastfeeding Education and Support Intervention on Timely Initiation and Exclusive Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Misra Abdulahi, Associate Professor, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BFESI
Record Dates: First submitted 2017-01-14; First posted 2017-01-25 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Breastfeeding, Exclusive; Nutrition Status
Keywords: Breastfeeding; Education and support; Ethiopia; Timely initiation of breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Education and Support (Experimental): Pregnant women in the intervention arm will receive breastfeeding education and support intervention for nine months starting in their third trimester
  Interventions: Behavioral: Breastfeeding Education and Support
- Usual or routine care (No Intervention): Pregnant women in the intervention arm will continue to receive the usual/routine care.

INTERVENTIONS:
Behavioral: Breastfeeding Education and Support — Women Development Army (WDA) leaders will function as peers for mothers in intervention group. There will be two visits during pregnancy and 8 visits postnatally. During pregnancy, WDA leaders will cover in detail the importance of EBF, feeding colostrum first, and discouraging prelacteal foods and encourage the mother to deliver at the nearby health center. During Postnatal visits, mothers will be observed positioning, attaching, and feeding the new-born, with appropriate feedback provided, solving any BF problems, encourage the mothers to continue exclusive breastfeeding for 6 months, emphasize nutrition for sufficient breast milk to breastfeed successfully and hands-on guidance only when necessary.
  Arms: Breastfeeding Education and Support

SUMMARY:
The purpose of this study is to develop and test Breastfeeding Education and Support Intervention for improving timely initiation and Exclusive Breastfeeding rate.

Infant mortality rates are still high in Ethiopia. Breastfeeding (BF) is regarded as the simplest and least expensive strategy for reduction of infant mortality rates. Ethiopia does not meet the international recommendation for exclusive breastfeeding (EBF) for the first six months of life. Community-based educational and support interventions provided prenatally and postnatally are effective in increasing BF rates. However, there is paucity of such information in Ethiopia.

DETAILED DESCRIPTION:
Sample size was calculated using Sample Size Calculator (SSC) a Windows based software package (93) with the following assumptions: to detect an increase in exclusive breastfeeding for 6 month from 52% to 72% (44), with 95% Confidence Intervals and 80% power, assuming an intra-cluster correlation coefficient of 0•1 from Ugandan study (94) for a cluster size of ten, it is calculated that we will need thirty six clusters. Adding 20% of the sample size for loss to follow-up, the final sample size is 432 pregnant women (216 in intervention, and 216 in control).

Standard operating procedure will be prepared and used for data collection. Data will be entered into Epi-data version 3.1 and analyzed using STATA version 12.0. Frequency distributions will be run to identify outliers. In relation to the trial hypotheses, intervention group will be compared to the routine education using intention to treat analysis. For the outcomes, proportions of women who initiated BF timely and who exclusively breastfed their babies at 72 hours and at 6 month will be compared using odds ratios derived using logistic regression between intervention and control groups. In all analyses, adjustment will be made for clustering at the zone level since randomization was done at cluster level rather than individual level. Generalized linear models will be used to calculate prevalence ratios (PR) for the categorical anthropometric outcomes. In the longitudinal analysis, the correlated nature of the data from the repeated measurements will be taken into account by adjusting for repeated measurements in the same individual as well as the above-mentioned design effect resulting from the cluster randomization. A linear mixed effects regression model will be used in the longitudinal analysis of z-scores with cluster as a random effect and the repeated measurements in each child accounted for through a first order autocorrelation structure. Least Squares Means (LSM) are reported at 3, 6 months, corresponding to the scheduled data collection visits.

ELIGIBILITY:
Inclusion Criteria:

During pregnancy

* pregnant women in the third trimester
* Live in the selected cluster and
* Have no plans to move away during the intervention period
* Without psychiatric illness
* Capable of giving informed consent and willing to be visited by supervisors and data collectors After delivery
* Singleton live birth with no severe malformation that could interfere with breastfeeding

Exclusion Criteria:

During pregnancy

* women with severe psychological illness which could interfere with consent and study participation
* Severely ill After delivery
* Severely ill or have clinical complications warranting hospitalization
* Stillbirth
* Infant death or maternal death
* Twin gestation
* Preterm birth (at <37 weeks gestation).

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-09-08 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | at six month
  Prevalence of exclusive breastfeeding (24-h recall) at month one, three and six in the intervention and control clusters.

SECONDARY OUTCOMES:
Timely initiation of breastfeeding | within 72 hours after delivery
  Prevalence of timely initiation of breastfeeding at month one in the intervention and control clusters.
Nutritional status | at months 3 and 6
  WHO Child Growth Standards (2006) will be used to estimate anthropometric status at months 3 and 6: weight-for-length z-scores (WLZ), length-for-age z-scores (LAZ) and weight-for-age z-scores (WAZ). Children who had WLZ below-2 (WLZ<-2) will be considered wasted, those with LAZ below -2(LAZ<-2) stunted, and those with WAZ below-2(WAZ<-2) underweight.
Knowledge towards breastfeeding | Baseline, at month 3 and 6
  Knowledge towards breastfeeding will be measured using the breastfeeding knowledge questionnaire after validating it.
Attitude towards breastfeeding | Baseline, at month 3 and 6
  Attitude towards breastfeeding will be measured using the Iowa Infant Feeding Attitude Scale (IIFAS) after validating it.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette H. Magnus, PhD, Study Director — University of Oslo; Atle Fretheim, PhD, Study Director — University of Oslo
Locations (1):
- Mana district, Jimma zone, Southwest Ethiopia, Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
participants flow, baseline characteristics, outcome measure statistical analysis

REFERENCES:
- [Derived] Abdulahi M, Fretheim A, Magnus JH. Effect of breastfeeding education and support intervention (BFESI) versus routine care on timely initiation and exclusive breastfeeding in Southwest Ethiopia: study protocol for a cluster randomized controlled trial. BMC Pediatr. 2018 Sep 26;18(1):313. doi: 10.1186/s12887-018-1278-5. PMID 30257661